CLINICAL TRIAL: NCT06723145
Title: Optimal PERioperative Antiplatelet Therapy Investigation ON Abdominal Surgery After Coronary Stent Implantation
Acronym: OPERATION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Hiroki Shiomi, Hiroki Shiomi MD, PhD, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0211; 24ek0210198h0001 (Other Grant/Funding Number: Japan Agency for Medical Research and Development)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Antiplatelet Agents; Perioperative Care
Keywords: antiplatelet agents; perioperative care; coroanry artery disease; abdominal disease; noncardiac surgery
MeSH Terms: interventions — Aspirin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin Continuation (Experimental): perioperative aspirin continuation
  Interventions: Drug: Aspirin
- Interruption of Antiplatelet Therapy (Active Comparator): Interruption of aspirin 5-7 days before surgery
  Interventions: Drug: Aspirin interruption

INTERVENTIONS:
Drug: Aspirin — perioperative aspirin continuation
  Other Names: Aspirin (drug)
  Arms: Aspirin Continuation
Drug: Aspirin interruption — Aspirin interruption 5-7 days before surgery
  Other Names: Aspirin interruption (drug)
  Arms: Interruption of Antiplatelet Therapy

SUMMARY:
The purpose of this study is to evaluate the impact of perioperative aspirin continuation on clinical outcomes in patients with a history of coronary stent implantation who are scheduled for abdominal surgery.

DETAILED DESCRIPTION:
PCI with coronary stent implantation is performed for a huge number of patients with coronary artery disease. Approximately 20% of these patients undergo non-cardiac surgery within three years after PCI. However, there is a scarcity of clinical evidence regarding the efficacy of perioperative aspirin continuation on cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of coronary stenting and scheduled for abdominal surgery
* Patients on a single antiplatelet agent

Exclusion Criteria:

* Patients on dual antiplatelet therapy (DAPT)
* Patients on anticoagulation therapy
* Patients with a history of stent thrombosis
* Patients with CHADS2 score >= 5
* Patients at extremely high risk of bleeding and unable to continue preoperative aspirin
* Patients incapable of consent, including those under 20 years of age
* Other patients for whom either discontinuation or continuation of antiplatelet agents is deemed inappropriate by the attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
a composite of death or myocardial infarction | 30 days
  the primary endpoint is defined as a composite of all-cause death or myocardial infarction (4th UDMI definition)

SECONDARY OUTCOMES:
Major bleeding (TIMI major/minor bleeding) | 30 days
  TIMI major/minor bleeding
Death/Myocardial Infarction (4th UDMI Definition)/Stroke | 30 days
  a composite of Death, Myocardial Infarction (4th UDMI Definition), or Stroke
Death/Myocardial Infarction (4th UDMI Definition)/Myocardial Injury (MINS) | 30 days
  a composite of Death, Myocardial Infarction (4th UDMI Definition), or Myocardial Injury (MINS)
Myocardial Infarction (4th UDMI Definition)/Myocardial Injury (MINS) | 30 days
  a composite of Myocardial Infarction (4th UDMI Definition), or Myocardial Injury (MINS)
Death/Myocardial Infarction (ARC-2 Definition)/Stroke | 30 days
  a composite of Death, Myocardial Infarction (ARC-2 Definition), orStroke
Death | 30 days
  all-cause death
Cardiovascular Death | 30 days
  cardac and vascular death
Myocardial Infarction (4th UDMI Definition) | 30 days
  Myocardial Infarction defined by 4th UDMI Definition
Myocardial Infarction (ARC-2 Definition) | 30 days
  Myocardial Infarction defined by ARC-2 Definition
Myocardial Infarction (SCAI Definition) | 30 days
  Myocardial Infarction defined by SCAI Definition
Myocardial Infarction (modified POISE-2 Definition) | 30 days
  Myocardial Infarction defined by modified POISE-2 Definition
Myocardial Injury (MINS) | 30 days
  Myocardial Injury (MINS) is defined as cardiac enzyme elevation without symptoms or ECG changes.
Stent Thrombosis (ARC Definition) | 30 days
  Stent thrombosis defined by ARC definition
Stroke | 30 days
  Sudden neurological disorder that persists for at least 24 hours and is caused by blockage of cerebral blood flow due to bleeding or ischemia.
Cerebral Infarction | 30 days
  Sudden neurological disorder that persists for at least 24 hours and is caused by infarction.
Cerebral Hemorrhage | 30 days
  Sudden neurological disorder that persists for at least 24 hours and is caused by cerebral bleeding.
Coronary Revascularization | 30 days
  PCI or CABG
Major Bleeding (BARC classification) | 30 days
  Major bleeding defined by BARC classification
Major Bleeding (modified POISE-2 classification) | 30 days
  Major bleeding defined by modified POISE-2 classification
Major Bleeding (GUSTO classification) | 30 days
  Major bleeding defined by GUSTO classification
Fatal Bleeding | 30 days
  Fatal bleeding within 30 days after abdominal surgery
Bleeding Volume During Non-Cardiac Surgery | 30 days
  bleeding volume during abdominal surgery
Transfusion | 30 days
  transfusion during and after surgery
Reoperation | 30 days
  any reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Shiomi, MD, PhD, Principal Investigator — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No